CLINICAL TRIAL: NCT03711916
Title: Pilot Study: Post-Operative Outcomes of Low Thermal Dissection vs. Traditional Electrosurgery for Mastectomy Breast Flap Creation With Immediate Breast Reconstruction
Brief Title: Post-Operative Outcomes of Low Thermal Dissection vs. Traditional Electrosurgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: Medtronic (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Device Feasibility
Other Study IDs: J1697; IRB00108493 (Other: JHM IRB)
Record Dates: First submitted 2018-10-17; First posted 2018-10-19 (Actual); Last update posted 2019-06-18 (Actual); Status verified 2019-06

CONDITIONS: Breast Cancer; Mastectomy; Perfusion; Complications; Hemostasis
Keywords: Breast cancer; Mastectomy; Perfusion; Hemostasis
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Breast flap creation with PlasmaBlade (Experimental): During participant's scheduled bilateral mastectomy, breast flap on one breast will be created using low thermal dissection device (PlasmaBlade) on one breast and standard Bovie cautery in the contralateral breast.
  Interventions: Device: PlasmaBlade 3.0S
- Breast flap creation with Bovie Cautery (No Intervention): During participant's scheduled bilateral mastectomy, breast flap will be created using standard Bovie cautery on the breast contralateral to the one that was created using PlasmaBlade.

INTERVENTIONS:
Device: PlasmaBlade 3.0S — PlasmaBlade (Medtronic) is approved by United States Food and Drug Administration (FDA) as a low thermal dissection device that has shown to be associated with effective cutting, and significantly lower temperature than traditional electrosurgical dissection devices.
  Arms: Breast flap creation with PlasmaBlade

SUMMARY:
Low thermal dissection devices have been introduced as a tool to improve surgical outcomes. PlasmaBlade, a low thermal dissection device, has shown to be associated with effective cutting, and significantly lower temperature than traditional electrosurgical dissection device. Thus, low thermal devices would improve flap perfusion by decreasing the thermal injury resulted by the dissection. Looking into the use of low thermal devices in cases of mastectomy and immediate breast reconstruction has not been documented. The aim of this study is to determine if there are clinical flap perfusion, surgical site drainage, and pain scores differences between mastectomy flaps created using low thermal dissection device and those done with the standard care of Bovie cautery in order to warrant a formal study.

DETAILED DESCRIPTION:
This is a single-blinded, randomized, controlled clinical trial comparing postoperative flap perfusion and surgical site drainage between patients randomized to breast flap creation by PlasmaBlade (low thermal dissection intervention) on one breast and by a Bovie cautery (Control) for the contralateral breast flap. Candidates will have elected to undergo bilateral post-mastectomy immediate breast reconstruction (IBR). Participants meeting inclusion criteria will be enrolled and baseline data collection completed prior to randomization and surgery.

Patients and the plastic surgeon will be blinded in regards to intervention randomization. Only the oncology surgeon has knowledge of which device used for each breast flap. However, after the plastic surgeon makes the assessment of the flap, he/she will be unblinded in order to complete the reconstruction procedure using the same dissection device on the same side it was used for in the mastectomy procedure. Patient-specific surgical details will be recorded intraoperatively. Following the surgery, post-operative flap perfusion will be recorded using SPY imaging system. Surgical site drainage will be measured until drainage removal. Post-operative pain (Visual Analog Scale for Pain) and the occurrence of adverse events will be recorded up until discharge and 30-days postoperative follow up visit.

ELIGIBILITY:
Inclusion Criteria:

* Women aged 18-75 years.
* Choose bilateral mastectomy followed by immediate breast reconstruction.
* Have no inflammatory breast cancers.
* Have not had radiotherapy before mastectomy.
* Understand the study purpose, requirements, and risks.
* Be able and willing to give informed consent.

Exclusion Criteria:

* Active connective tissue disease.
* History of, or plan to undergo irradiation of the breasts.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Only enrolling women undergoing bilateral mastectomy
Enrollment: 20 (Actual)
Dates: Start 2017-03-17 (Actual); Primary Completion 2018-10-24 (Actual); Study Completion 2018-12-03 (Actual)

PRIMARY OUTCOMES:
Perfusion | Day of Surgery
  Plastic surgeon objectively assesses degree of perfusion with the SPY Perfusion Assessment system (intra-operative fluorescence imaging system). Plastic surgeon describes perfusion as Left better than Right, Right better than Left, or both sides equally perfused.

SECONDARY OUTCOMES:
Drainage | Up to 14 days post-operatively.
  Patient records amount of drainage (in cc's) from each drain until drain is removed by plastic surgeon.
Pain Scores | Days 1,2,3,7,30 Post-operatively
  Patient records pains scores using Visual Analog Scale (10cm long line upon which patients indicates level of pain)for each side at Day 1, 2, 3, 7, and 30. Scores range from 0-10. Score of 0 corresponds with 0 cm on the line and 10 corresponds with 10cm on the line. 0 indicates no pain and 10 indicates most severe pain.

CONTACTS AND LOCATIONS:
Overall Officials: Mehran Habibi, MD, Principal Investigator — Johns Hopkins Medicine Department of Surgery; Gedge D Rosson, MD, Principal Investigator — Johns Hopkins Medicine Department of Plastic, Reconstructive & Maxillofacial Surgery
Locations (2):
- United States (2):
  - Bayview Medical Center, Baltimore, Maryland
  - Johns Hopkins Hospital Outpatient Center, Baltimore, Maryland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Habibi M, Prasath V, Dembinski R, Sacks JM, Rosson GD, Sebai ME, Mirkhaef S, Bello RJ, Siotos C, Broderick KP. Comparison of mastectomy and breast reconstruction outcomes using low thermal dissection versus traditional electrocautery: a blinded randomized trial. Breast Cancer Res Treat. 2021 Jul;188(1):101-106. doi: 10.1007/s10549-021-06177-9. Epub 2021 Mar 19. PMID 33742323